CLINICAL TRIAL: NCT06361706
Title: Desenvolupament i Avaluació de l'Experiència en Realitat Virtual en la Prova Pilot Per a Pacients Amb Dolor Crònic i Sensibilització Central Als Centres d'Atenció Primària de Badalona Serveis Assistencials
Brief Title: VR-Enhanced Psychoeducation for Chronic Pain: A Primary Care Pilot Study
Acronym: REDOCVR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Badalona Serveis Assistencials (Other)
Collaborators: Department of Health, Generalitat de Catalunya (Other Government)
Responsible Party: Principal Investigator, Jose Ferrer Costa, Clinical Researcher at the Innovation and Projects department, Badalona Serveis Assistencials
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 24/047-P
Record Dates: First submitted 2024-04-07; First posted 2024-04-12 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-05

CONDITIONS: Chronic Pain; Central Sensitization
Keywords: chronic pain; central sensitization; virtual reality; patient education as a topic; pain management; behavioral therapy; digital health; primary health care
MeSH Terms: conditions — Chronic Pain; Agnosia

STUDY DESIGN:
Intervention Model Description: The REDOCVR study utilizes a Single-Group Interventional Model, where all participants receive the same VR-enhanced psychoeducational intervention for chronic pain management. This model facilitates a focused evaluation of VR's effectiveness and usability within a structured psychoeducational framework, allowing for direct assessment of participant experiences and outcomes.
Masking Description: The statisticians and researchers involved in data analysis will be masked to the identity of participants, using a random code for each participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VR-Enhanced Chronic Pain Management Program (Experimental): Participants in this arm will undergo a comprehensive psychoeducational program tailored for chronic pain and central sensitization management, significantly enhanced with Virtual Reality (VR) experiences.
  Interventions: Behavioral: VR-Enhanced Psychoeducational Program for Chronic Pain

INTERVENTIONS:
Behavioral: VR-Enhanced Psychoeducational Program for Chronic Pain — Participants undergo eight weekly sessions that include VR to learn pain physiology, mindfulness, and self-management techniques. Each session is 90 minutes, with 15-20 minutes of VR activities designed to complement the educational content. Activities simulate pain management exercises and mindfulness meditation. The program, led by pain management and VR specialists, aims to improve pain management skills, emotional well-being, and quality of life.

SUMMARY:
This pilot study aims to evaluate the integration of virtual reality (VR) with a psychoeducational program for individuals experiencing chronic pain and central sensitization. Chronic pain significantly hampers daily life, and the condition of central sensitization intensifies this challenge by making the pain more acute. Our research is grounded in the hypothesis that VR, when used to complement conventional psychoeducational methods, can enhance engagement and understanding of pain management strategies, thus potentially improving patient outcomes.

Key objectives and related measured variables include:

Usability and Feasibility: Evaluated through the System Usability Scale (SUS) responses from both participants and healthcare professionals, assessing the ease of use and integration of VR into the psychoeducational program.

Participant Engagement and Program Adherence: Determined by participants' satisfaction with the VR system, using Likert scale questionnaires, and tracked through session attendance and program completion rates.

Impact on Chronic Pain Management and Emotional Well-being: Assessed through changes in the Warwick-Edinburgh Mental Well-being Scale (WEMWBS), and the Hospital Anxiety and Depression Scale (HADS) collected at baseline, post-intervention, and 4-8 weeks follow-up Self-management of Chronic Pain: Monitored through the Central Sensitization Inventory (CSI) and changes in patient functionality and mobility using the EuroQol-5D-5L scale, measured at baseline, post-intervention, and 4-8 weeks follow-up.

Healthcare Professionals' Perceptions: Investigated using SUS scores and qualitative feedback on the applicability and benefits of VR in clinical practice for chronic pain management.

Participants will complete eight 90-minute sessions, engaging with VR to supplement the program's content. This approach aims to provide immersive experiences that deepen the understanding and management of chronic pain. Participant feedback on the VR experience, alongside observed changes in pain management and overall well-being, will be critically examined.

By targeting individuals suffering from chronic pain, this research aims to offer healthcare professionals an innovative tool for enhancing pain management strategies. Integrating VR into psychoeducational content, the study seeks to promote more engaging and effective learning experiences, potentially leading to improved outcomes in chronic pain management.

DETAILED DESCRIPTION:
The REDOCVR study is an innovative initiative to evaluate the adjunctive use of Virtual Reality (VR) within a psychoeducational framework for managing chronic pain and central sensitization. This initiative aims to harness the immersive potential of VR to enhance traditional psychoeducational strategies, thereby providing a more engaging and impactful patient experience.

Study Design Overview:

The study is structured as a prospective, non-randomized pilot intervention spanning September 2023 to December 2025 across select Primary Care Centers within Badalona Serveis Assistencials. Targeting adults with chronic pain, the intervention seeks to determine the feasibility, usability, and preliminary efficacy of incorporating VR into pain management protocols.

Recruitment and Selection Process Initial Information: The Primary Care Team is informed about the study and introduces it to potential participants that they identifiy in their daily clinical work, who are then scheduled for an evaluation through the centers electronic system.

Selection Procedure: Interested candidates are contacted via phone for further selection through a face-to-face recruitment visit, assessing eligibility by the Inclusion and Exclusion Criteria and collecting informed consent along with baseline data.

Data Collection and Analysis Specifics:

Data will be meticulously collected on paper before being digitized for analysis, ensuring a robust process for capturing and analyzing participant responses, feedback, and outcomes. This process underscores the study's commitment to methodological rigor and data integrity.

Ethical Considerations: Detailed information on informed consent, data management, privacy, and confidentiality will be addressed in the ethical considerations section.

Innovative Intervention Approach:

Participants are introduced to VR as a tool for understanding and managing their condition, with sessions designed to align VR experiences with educational content. The program includes 8 weekly sessions, each lasting 90 minutes, with VR experiences embedded into the curriculum to reinforce learning objectives and engage participants in their care process actively.

Technological and Methodological Framework:

The intervention leverages Oculus Quest 2 headsets, chosen for their standalone capability and immersive quality. Custom content developed using Unity software focuses on mindfulness, pain education, and self-management techniques, ensuring that VR sessions are directly relevant to participants' learning and therapeutic goals.

Overview of Sessions The intervention framework consists of 8 weekly, 90-minute sessions conducted in session rooms within healthcare centers. Each session incorporates a dedicated 15-20 minute segment for VR experiences designed to complement the session's theme and objectives.

Recruitment Visit A 30-minute recruitment visit initiates the study process, involving eligibility assessment through anamnesis, detailing the study's scope, and gathering informed consent from participants.

Session Breakdown

1. Introduction to VR Begins with an overview presented by healthcare professionals, followed by an introduction to VR technology, including a practical demonstration to acquaint patients with VR, capped with a 15-minute mindfulness technique using VR.
2. Pain Neurophysiology and Self-management Techniques Focuses on explaining the neurophysiology of pain and introducing pain self-management techniques, including habit changes. Features an educational video to deepen the acquired knowledge.
3. Psychological Aspects of Pain Concentrates on the psychological dimensions of pain, including the gate control theory. Utilizes 360-degree VR videos, controlled by a psychologist with a tablet, explaining techniques for pain awareness and acceptance.

4 & 6: Reeducation of the Central Nervous System (CNS) Through Physical Activity Engages patients in CNS reeducation activities using interactive VR games designed to encourage physical activity in a fun and engaging manner, overseen by a physiotherapist.

5: Psychological Aspects of Pain - Emotions and Thoughts Addresses emotions and thoughts associated with chronic pain through an educational VR session on emotional management techniques.

7: Emotions and Self-esteem Focuses on acceptance, self-esteem, and emotion management, incorporating a VR educational session on compassionate acceptance techniques.

8: Farewell A closing session that reviews covered content and concludes with a final VR session on attentive breathing techniques for relaxation and skill consolidation.

Expected Outcomes and Contributions:

Through a detailed exploration of VR's role in psychoeducation for chronic pain, the REDOCVR study aims to provide valuable insights into how digital health innovations can enhance traditional therapeutic modalities. The findings are anticipated to inform future interventions, guide clinical practice, and contribute to the broader dialogue on integrating technology into patient care.

ELIGIBILITY:
Inclusion Criteria:

* Patients experiencing chronic pain with elements of central sensitization, emotional discomfort related to pain, kinesiophobia, or inadequate response to prescribed treatments.
* Patients aged 18 years or older assigned to the assigned to Badalona Serveis Assistnecials´ Primary Care.
* Patients capable of providing consent to participate in the study, signing the informed consent form, and responding to the variable-related questions.

Exclusion Criteria:

* Patients with acute pain (less than 3 months)
* Diagnosis of systemic diseases or severe mental disorders, cognitive impairment, vertigo, epilepsy, or significant visual/auditory impairments that prevent the use of VR headsets.

Withdrawal Criteria:

- Presence of VR-related side effects or patient's decision to withdraw.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-12-04 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Participant Satisfaction with the VR-enhanced Psychoeducational Program as measured by the Participants Satisfaction Questionnaire | Immediately after the last intervention session (within 30 minutes of completing the 8th session)
  The Participant Satisfaction Questionnaire assesses with 10 itens various aspects of the VR-enhanced psychoeducational program, including content relevance, VR experience, and perceived benefits in managing chronic pain. This questionnaire uses a Likert scale for responses, providing a quantitative measure of participant satisfaction. The questionnaire's design allows for a comprehensive evaluation of the program's impact on participants, with higher scores indicating greater satisfaction.
Participants´ System Usability and VR Headset Comfort as assessed by the SUS for participants | Immediately after the last intervention session (within 30 minutes of completing the 8th session)
  The SUS is a two-part Likert Scale with options ranging from "Strongly disagree" to "I quite agree," designed to evaluate both the system's usability and the comfort of the VR headset used. Participants will respond to 16 statements, with 8 focused on system usability and 8 on headset comfort. Statements are rated on a scale from 1 to 5. For usability, positive experiences are reflected by statements 1, 3, 4, 6, and 7, while for headset comfort, statements assess aspects like weight, ease of use, and physical discomfort. The overall SUS score is calculated to assess usability and comfort, with higher scores indicating better usability and comfort levels.
Professionals System Usability as measured by the SUS for Professionals | Immediately after the last intervention session (within 30 minutes of completing the 8th session)
  The SUS for Professionals is designed to evaluate healthcare professionals' perceptions of the VR system's usability within the clinical setting for this educational program. This assessment uses a Likert Scale from "Strongly disagree" to "I quite agree," focusing on ease of use, integration into practice, and the system's effectiveness in enhancing patient care. Higher scores on the SUS for Professionals indicate a positive assessment of the system's usability and potential impact on patient treatment.

SECONDARY OUTCOMES:
Mental Well-being as assessed by the WEMWBS-7 | Baseline and immediately after the last intervention session (within 30 minutes of completing the 8th session)
  The 7-item Warwick-Edinburgh Mental Well-being Scale (WEMWBS-7) is a concise version designed to efficiently assess mental well-being, focusing predominantly on functioning aspects. It is characterized by better scaling properties, enhancing the precision of measuring differences in scores. It has been demonstrated to be responsive to change in clinical populations undergoing psychotherapy at both group and individual levels. The minimal detectable change at the individual level is calculated as 1 or 3 points, with total scores requiring transformation according to a provided table. This scale is chosen for its brevity and focus on functioning, making it particularly suited for evaluations where time is constrained but a precise and responsive measure of mental well-being is needed.
Anxiety and Depression Severity as measured by the HADS | Baseline and immediately after the last intervention session (within 30 minutes of completing the 8th session)
  The Hospital Anxiety and Depression Scale (HADS) is a self-administered instrument consisting of 14 items divided into two subscales: one for anxiety and one for depression, with interspersed items. It focuses on anhedonia as a core aspect of the depression subscale, a primary symptom distinguishing depression from anxiety. Items are scored on a 4-point Likert frequency scale (0-3), with total scores ranging from 0 to 21 for each subscale. Higher scores indicate greater symptom severity. Scores above eleven suggest a definitive "case" of anxiety or depression, while scores above eight are considered "probable cases." The scale's internal consistency for the Spanish population in a fibromyalgia study was α=.83 for anxiety and α=.87 for depression.
Central Sensitization as measured by the CSI | Baseline and immediately after the last intervention session (within 30 minutes of completing the 8th session)
  The Central Sensitization Inventory (CSI) is utilized to assess the extent of central sensitization symptoms in participants. It comprises questions rated on a 5-point scale, from 0 ("never") to 4 ("always"), with the total score achievable being 100. This summed response quantifies the level of self-reported symptomology related to central sensitization. Higher CSI scores indicate greater symptom severity, with a score exceeding 40 suggesting the presence of central sensitization. This measure is critical for identifying participants experiencing heightened sensitivity to pain, a key factor in chronic pain syndromes, and assessing the effectiveness of interventions aimed at managing these symptoms.
Changes in Functionality and Mobility as assessed by the EuroQol-5D-5L Scale | Baseline and immediately after the last intervention session (within 30 minutes of completing the 8th session)
  The EuroQol-5D-5L scale measures changes in participants' functionality and mobility. This assessment covers five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, with a scoring system that highlights the degree of difficulty in each area. Improvements are indicated by lower scores in dimensions related to pain/discomfort and better scores in mobility and self-care.
Adherence to the VR-enhanced Psychoeducational Program as indicated by session attendance and program completion rates | After the last intervention session, up to 16 weeks
  Program adherence is measured by tracking participants' attendance at the sessions and their completion of the entire VR-enhanced psychoeducational program. High attendance and completion rates are indicators of the program's acceptability and participants' engagement with the VR intervention.

OTHER OUTCOMES:
Participant Feedback as recorded on the Participant Comment Sheet | Immediately at the end of each session
  The Participant Comment Sheet is designed to capture immediate, qualitative feedback from participants at the end of each VR-enhanced psychoeducational session. This open-ended feedback mechanism allows participants to express their thoughts, experiences, and suggestions regarding the session they just completed. The comments provide valuable insights into the program's reception, areas for improvement, and the overall impact from the participant's perspective. Collecting this data after each session enables ongoing evaluation and potential adjustment of the program based on participant feedback, enhancing the relevance and effectiveness of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Ferrer Costa, MD, Principal Investigator — Badalona Serveis Assistencials
Locations (4):
- Spain (4):
  - Primary Care Progrès-Raval, Badalona, Barcelona
  - Primary Care Center Apenins-Montigalà, Badalona, Barcelona
  - Primary Care Center Morera-Pomar, Badalona, Barcelona
  - CAP Montgat- Dr Jardi, Montgat, Barcelona

IPD SHARING:
Plan to Share IPD: Yes
In our study, outcome data initially collected on paper are manually entered into Excel sheets, creating a digitized dataset that reflects the raw results of the research. This digitization process is conducted with precision to ensure accuracy and reliability of the data. The digitalized data are then coded and stored securely within the BSA intranet, in a protected digital folder accessible only to authorized personnel.
  Given the manual transcription and internal storage of these data, our plan to share Individual Participant Data (IPD) includes specific steps tailored to maintain data integrity, confidentiality, and compliance with ethical standards:
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The digitized IPD will be made available to approved researchers starting 12 months after the publication of the main study results. This window allows sufficient time for the meticulous preparation of the data for external use. The data will be accessible for a period of up to 3 years, during which requests for access can be submitted and reviewed.
Access Criteria: Access to IPD will be granted to researchers submitting scientifically valid proposals that align with ethical guidelines. A review committee will evaluate proposals based on their objectives, methodology, and compliance with data protection standards. Successful applicants will sign a data use agreement detailing secure data handling and confidentiality requirements. Instructions for secure data access, including anonymization protocols and secure transfer methods, will be provided to approved researchers. Data will be accessible via a secure platform within the BSA intranet, ensuring data integrity and participant privacy are maintained.

REFERENCES:
- [Background] Brown CA, Jones AK. Psychobiological correlates of improved mental health in patients with musculoskeletal pain after a mindfulness-based pain management program. Clin J Pain. 2013 Mar;29(3):233-44. doi: 10.1097/AJP.0b013e31824c5d9f. PMID 22874090
- [Background] Grossman P, Tiefenthaler-Gilmer U, Raysz A, Kesper U. Mindfulness training as an intervention for fibromyalgia: evidence of postintervention and 3-year follow-up benefits in well-being. Psychother Psychosom. 2007;76(4):226-33. doi: 10.1159/000101501. PMID 17570961
- [Background] Ma J, Zhao D, Xu N, Yang J. The effectiveness of immersive virtual reality (VR) based mindfulness training on improvement mental-health in adults: A narrative systematic review. Explore (NY). 2023 May-Jun;19(3):310-318. doi: 10.1016/j.explore.2022.08.001. Epub 2022 Aug 5. PMID 36002363
- [Background] Yang H, Cai M, Diao Y, Liu R, Liu L, Xiang Q. How does interactive virtual reality enhance learning outcomes via emotional experiences? A structural equation modeling approach. Front Psychol. 2023 Jan 6;13:1081372. doi: 10.3389/fpsyg.2022.1081372. eCollection 2022. PMID 36687987
- [Background] Moro C, Stromberga Z, Raikos A, Stirling A. The effectiveness of virtual and augmented reality in health sciences and medical anatomy. Anat Sci Educ. 2017 Nov;10(6):549-559. doi: 10.1002/ase.1696. Epub 2017 Apr 17. PMID 28419750
- [Background] Barteit S, Lanfermann L, Barnighausen T, Neuhann F, Beiersmann C. Augmented, Mixed, and Virtual Reality-Based Head-Mounted Devices for Medical Education: Systematic Review. JMIR Serious Games. 2021 Jul 8;9(3):e29080. doi: 10.2196/29080. PMID 34255668
- [Background] Pascual K, Fredman A, Naum A, Patil C, Sikka N. Should Mindfulness for Health Care Workers Go Virtual? A Mindfulness-Based Intervention Using Virtual Reality and Heart Rate Variability in the Emergency Department. Workplace Health Saf. 2023 Apr;71(4):188-194. doi: 10.1177/21650799221123258. Epub 2022 Nov 14. PMID 36377263
- [Background] Meese MM, O'Hagan EC, Chang TP. Healthcare Provider Stress and Virtual Reality Simulation: A Scoping Review. Simul Healthc. 2021 Aug 1;16(4):268-274. doi: 10.1097/SIH.0000000000000484. PMID 32890319
- [Background] Tack C. Virtual reality and chronic low back pain. Disabil Rehabil Assist Technol. 2021 Aug;16(6):637-645. doi: 10.1080/17483107.2019.1688399. Epub 2019 Nov 20. PMID 31746250
- [Background] Goudman L, Jansen J, Billot M, Vets N, De Smedt A, Roulaud M, Rigoard P, Moens M. Virtual Reality Applications in Chronic Pain Management: Systematic Review and Meta-analysis. JMIR Serious Games. 2022 May 10;10(2):e34402. doi: 10.2196/34402. PMID 35536641
- [Background] Ummels D, Cnockaert E, Timmers I, den Hollander M, Smeets R. Use of Virtual Reality in Interdisciplinary Multimodal Pain Treatment With Insights From Health Care Professionals and Patients: Action Research Study. JMIR Rehabil Assist Technol. 2023 Nov 10;10:e47541. doi: 10.2196/47541. PMID 37948109
- [Background] de Vries FS, van Dongen RTM, Bertens D. Pain education and pain management skills in virtual reality in the treatment of chronic low back pain: A multiple baseline single-case experimental design. Behav Res Ther. 2023 Mar;162:104257. doi: 10.1016/j.brat.2023.104257. Epub 2023 Jan 18. PMID 36731183
- [Background] Brown L, DiCenso-Fleming T, Ensign T, Boyd AJ, Monaghan G, Binder DS. Chronic pain education delivered with a virtual reality headset in outpatient physical therapy clinics: a multi-site exploratory trial. Am J Transl Res. 2023 May 15;15(5):3500-3510. eCollection 2023. PMID 37303618